CLINICAL TRIAL: NCT03060993
Title: Effect of Inhaled Vaporized Cannabis on Pulmonary Function, Breathlessness and Exercise Tolerance in Symptomatic Patients With Advanced Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: CAN BREATHE in COPD Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Dennis Jensen, Ph.D., Assistant Professor, McGill University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNBS001
Record Dates: First submitted 2017-02-11; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Breathlessness; Exercise Intolerance
Keywords: Cannabis; Marijuana
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): 35 mg of tetrahydrocannabinol/cannabidiol (LT1.0/LT1.0 %) in vaporized form. Placebo will be vaporized using the Volcano Medic vaporizer. Total volume of vapour administered to each patient will be 5.5 L.
  Interventions: Drug: Placebo
- Cannabis (Active Comparator): 35 mg of cannabis (tetrahydrocannabinol/cannabidiol; 18.0/LT1.0 %) in vaporized form. THC/CBD will be vaporized using the Volcano Medic vaporizer. Total volume of vapour administered to each patient will be 5.5 L.
  Interventions: Drug: Cannabis

INTERVENTIONS:
Drug: Cannabis — Patients will be administered cannabis (THC/CBD) in vaporized form.
  Arms: Cannabis
Drug: Placebo — Patients will be administered placebo (cannabis stripped of cannabinoids) in vaporized form.
  Arms: Placebo

SUMMARY:
A growing body of physiological evidence now exists to support a potential role for inhaled cannabis in the medical management of adults with chronic obstructive pulmonary disease (COPD), particularly as it may related to improving pulmonary function, alleviating the symptom of breathlessness and improving exercise endurance. The purpose of this randomized double-blind crossover trials is to evaluate the efficacy and physiological mechanism(s) of action of inhaled vaporized cannabis targeted to relief of physical activity-related breathlessness and exercise endurance in symptomatic patients with severe-to-very severe COPD.

ELIGIBILITY:
Inclusion Criteria:

* GOLD stage III or IV COPD (i.e., post-β2-agonist FEV1 of 50% predicted or less)
* Self-reported cigarette smoking history ≥10 pack yrs
* Currently taking long-acting beta-2 agonists and long-acting antimuscarinic agents (LABA/LAMAs) with or without an inhaled corticosteroid
* Willing to abstain from cannabis smoking for ≥15 days prior to study participation (if applicable)
* Willing to abstain from non-study related cannabis smoking throughout the study period (if applicable)
* No change in medication dosage or frequency of administration, with no exacerbations or hospitalizations in the preceding 4 weeks

Exclusion Criteria:

* Presence of active and/or uncontrolled cardiopulmonary and/or musculoskeletal disease other than COPD that could contribute to breathlessness and exercise intolerance
* Hepatic or renal impairment
* Psychiatric history (other than depression and/or anxiety)
* History of epilepsy or convulsions;
* Lung cancer
* History of sensitivity to cannabis
* Use of levodopa, sildenafil and/or fentanyl
* Use of ketoconazole
* Use of regular high dose opioids (i.e., 30 mg of oral morphine equivalents/day)
* Known or suspected history of addiction/substance abuse based on CAGE-AID and SISAP scores (*note, patients may be recruited if they have a history of smoking cannabis)
* Positive urine toxicology for cannabinoids on screening
* Positive pregnancy urine test
* Subject cannot arrange to be accompanied home by a family member and/or friend during each treatment visit.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2017-03-01 (Estimated); Primary Completion 2018-01-01 (Estimated); Study Completion 2018-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes in intensity ratings of perceived breathlessness at isotime during cycle exercise testing. | Participants will be followed until all study visits are complete, an expected average of 4 weeks
  Patients will be required to rate the intensity of their breathlessness using Borg's modified 0-10 category ratio scale every 2-minutes during cycle exercise testing.
Changes in cycle exercise endurance time. | Participants will be followed until all study visits are complete, an expected average of 4 weeks
  Exercise endurance time will be defined as the duration of loaded pedaling during the constant-load cycle exercise testing performed at 75% of peak incremental power output.

SECONDARY OUTCOMES:
Changes in Spirometry | Participants will be followed until all study visits are complete, an expected average of 4 weeks
  Spirometry will be performed before and 5-min after treatment administration
Changes in Impulse oscillometry | Participants will be followed until all study visits are complete, an expected average of 4 weeks
  Impulse oscillometry will be performed before and 10-min after treatment administration
Changes in Physiological responses during exercise. | Participants will be followed until all study visits are complete, an expected average of 4 weeks
  Gas exchange, cardiovascular and breathing pattern variables will be collected breath-by-breath and averaged in 30-sec epochs during incremental and constant-load cycle exercise tests.
Plasma cannabinoid levels. | Participants will be followed until all study visits are complete, an expected average of 4 weeks
  Venous blood samples for the determination of circulating levels of cannabinoids will be collected before and 2-, 30-, 75-, and 180-min after vaporization
Psychoactive effects. | Participants will be followed until all study visits are complete, an expected average of 4 weeks
  Psychoactive effects of cannabis will be evaluated during each treatment visit using 100-mm visual analogue scale (VAS). Psychoactive effects will be evaluated before and 45-min after treatment administration.
Mood effects. | Participants will be followed until all study visits are complete, an expected average of 4 weeks
  Mood effects of cannabis will be evaluated during each treatment visit using 100-mm visual analogue scale (VAS). Mood effects will be evaluated before and 45-min after treatment administration.
Cognitive effects. | Participants will be followed until all study visits are complete, an expected average of 4 weeks
  Cognitive effects will be measured during each treatment visit using the mini-mental state exam. The mini-mental state exam will be administered before and 45-min after treatment administration

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Jensen, Ph.D., Principal Investigator — McGill University
Locations (1):
- McConnell Centre for Innovative Medicine, Research Institute of the McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdallah SJ, Smith BM, Ware MA, Moore M, Li PZ, Bourbeau J, Jensen D. Effect of Vaporized Cannabis on Exertional Breathlessness and Exercise Endurance in Advanced Chronic Obstructive Pulmonary Disease. A Randomized Controlled Trial. Ann Am Thorac Soc. 2018 Oct;15(10):1146-1158. doi: 10.1513/AnnalsATS.201803-198OC. PMID 30049223
- See also: Clinical Exercise & Respiratory Physiology Laboratory (CERPL) of McGill University — http://www.mcgill.ca/cerpl/